CLINICAL TRIAL: NCT01674842
Title: A Phase I Dose-Escalation Study of Cisplatin and Radiation Therapy for Patients With Triple Negative Breast Cancer
Brief Title: Cisplatin + RT for Triple Negative Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jennifer Bellon, Principal Invstigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-283
Record Dates: First submitted 2012-08-23; First posted 2012-08-29 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer
Keywords: Triple negative; Stage II; Stage III
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cisplatin + Radiation Therapy (Experimental): Cisplatin concurrently with radiation therapy
  Interventions: Radiation: Radiation Therapy; Drug: Cisplatin

INTERVENTIONS:
Radiation: Radiation Therapy — Once daily, Monday - Friday for six weeks
Drug: Cisplatin — Intravenously, once weekly for six weeks
  Other Names: CDDP

SUMMARY:
This is a Phase I dose escalation study of cisplatin and concurrent radiation in patients with ER negative, PR negative and HER2 negative breast cancer who have undergone breast-conserving surgery or mastectomy.

Primary objective: To assess the safety, tolerability, and maximum tolerated dose (MTD) of cisplatin when given concurrently with radiation therapy for participants with Stage II or III breast cancer who have undergone breast conserving surgery or mastectomy

DETAILED DESCRIPTION:
This is a phase I dose escalation study of cisplatin and radiation to determine the toxicity of this combined treatment and establish an MTD.

ELIGIBILITY:
Inclusion Criteria:

* Primary tumor is triple negative breast cancer
* Breast-conserving surgery or mastectomy with surgical excision of all gross disease with negative surgical margins
* Pathologic or clinical stage II or III disease
* At least 3 week interval from last chemotherapy administration/breast surgery to radiation (no more than 8 weeks)

Exclusion Criteria:

* Pregnant or breastfeeding
* Prior radiation to breast or ipsilateral regional nodes
* Ongoing therapy with other investigational agents
* Hormonal therapy
* Significant co-morbidity
* Pathologic complete response following preoperative chemotherapy
* Biopsy proven metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-10; Primary Completion 2018-08 (Actual); Study Completion 2021-06-08 (Actual)

PRIMARY OUTCOMES:
Safety of Cisplatin w/ Radiation | 2 years
  To determine the maximum tolerated dose of cisplatin when given concurrently with radiation therapy for participants with Stage II or III breast cancer who have undergone breast conserving surgery or mastectomy.

SECONDARY OUTCOMES:
Local recurrence at 5 years | 5 years
  To assess local recurrence at 5-years in participants receiving cisplatin concurrently with radiation, as compared with historic controls receiving radiation without concurrent chemotherapy.
Long term toxicity | 2 years
  To assess long-term toxicity in participants receiving cisplatin concurrently with radiation

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer R Bellon, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber at Milford, Milford, Massachusetts
  - Dana Farber at South Shore Hospital, Weymouth, Massachusetts

REFERENCES:
- [Derived] Bellon JR, Chen YH, Rees R, Taghian AG, Wong JS, Punglia RS, Shiloh RY, Warren LEG, Krishnan MS, Phillips J, Pretz J, Jimenez R, Macausland S, Pashtan I, Andrews C, Isakoff SJ, Winer EP, Tolaney SM. A Phase 1 Dose-Escalation Trial of Radiation Therapy and Concurrent Cisplatin for Stage II and III Triple-Negative Breast Cancer. Int J Radiat Oncol Biol Phys. 2021 Sep 1;111(1):45-52. doi: 10.1016/j.ijrobp.2021.03.002. Epub 2021 Mar 10. PMID 33713742